CLINICAL TRIAL: NCT04030507
Title: Screening Magnetic Resonance Imaging of the Brain in Patients With Metastatic Breast Cancer Managed With First/Second Line Chemotherapy or Inflammatory Breast Cancer Managed With Definitive Intent: A Prospective Study
Brief Title: Screening Magnetic Resonance Imaging of the Brain in Patients With Breast Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Conquer Cancer Foundation (Other)
Responsible Party: Principal Investigator, Ayal Aizer, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 19-066
Record Dates: First submitted 2019-07-19; First posted 2019-07-24 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer; HER2-positive Breast Cancer; Triple Negative Breast Cancer; Hormone Receptor Positive Malignant Neoplasm of Breast; Inflammatory Breast Cancer; Metastatic Breast Cancer
Keywords: Breast Cancer; HER2-positive Breast Cancer; Triple Negative Breast Cancer; Hormone Receptor Positive Malignant Neoplasm of Breast; Inflammatory Breast Cancer; Metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms; Triple Negative Breast Neoplasms; Inflammatory Breast Neoplasms | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Inflammatory Breast Cancer Managed with Curative Intent (Experimental): * Patients will receive an initial screening magnetic resonance imaging (MRI) of the brain
  * If no evidence of intracranial involvement is identified, additional screening MRIs of the brain every six months for two years and at initial systemic progression.
  Interventions: Device: MRI
- HR+ or HER2+ Metastatic Breast Cancer - Screening Arm (Experimental): * An initial MRI screening will be conducted
  * If negative, patients will receive a second MRI of the brain at first systemic progression after study entry
  Interventions: Device: MRI
- HR+ or HER2+ Metastatic Breast Cancer - No Screening Arm (No Intervention): No initial MRI screening will be conducted
- Triple Negative Breast Cancer (Experimental): * An initial MRI screening will be conducted
  * If negative, patients will receive a second MRI of the brain at first systemic progression after study entry
  Interventions: Device: MRI

INTERVENTIONS:
Device: MRI — MRI (which stands for magnetic resonance imaging) provide imaging of the brain which help look for brain metastases (spread of the breast cancer to the brain).
  Other Names: Magnetic Resonance Imaging
  Arms: HR+ or HER2+ Metastatic Breast Cancer - Screening Arm; Inflammatory Breast Cancer Managed with Curative Intent; Triple Negative Breast Cancer

SUMMARY:
This research study is studying the usefulness of magnetic resonance imaging (MRI) to screen for brain metastases (spread of the breast cancer to the brain).

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials examine the safety and effectiveness of an investigational intervention, in this case magnetic resonance imaging (MRI) of the brain, to learn whether it is helpful in managing a specific disease.

In this research study, the investigators are utilizing screening MRIs of the brain to evaluate breast cancer patients for metastases to the brain. The investigators hope to understand whether screening MRIs of the brain can be implemented into the standard of care to earlier detect brain metastases in a population where screening MRIs of the brain are not currently recommended or systematically performed.

This trial will contain 4 cohorts:

1. Those with triple negative breast cancer (TNBC) will undergo screening MRI of the brain as part of a single arm, non-comparative study

2+3. Those with hormone receptor positive/(human epidermal growth factor receptor 2 (HER2) negative (HR+/HER2-) and HER2 positive (HER2+) subtypes will be randomized to receipt of screening MRI of the brain or no screening MRI of the brain to definitively test the value of MRI screening.

4. Patients with inflammatory breast cancer being treated with curative intent will undergo screening MRI of the brain as part of a single arm, non-comparative study.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed breast cancer with pathologic assessment of estrogen receptor (ER), progesterone receptor (PR), and (human epidermal growth factor receptor 2 (HER2) status. If subtype has changed over the course of a patient's disease, the treating clinician and/or study PI is responsible for selecting the subtype that most likely reflects the preponderance of oncologic disease at the time of enrollment.
* Participants must have radiographic evidence of extracranial, distant metastases or unresectable, locally recurrent breast cancer and be initiating (within 8 weeks of registration) first-line or second-line chemotherapy for their metastatic/recurrent disease OR inflammatory breast cancer being managed with curative intent within six months of diagnosis.
* Participants must be age 18 years or older.
* Participants must have a life expectancy of greater than 12 weeks.
* Participants must be willing to undergo study procedures.
* The effects of gadolinium / other magnetic resonance imaging (MRI)-based contrast agents on the developing human fetus are unknown. For this reason, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately.
* Participants must possess the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Participants who have a contraindication to MRI (e.g. noncompatible implanted metallic device for which MRI is absolutely contraindicated).
* Participants who have chronic kidney disease stage IV-V or end stage renal disease.
* Participants with a history of anaphylactic reactions to gadolinium.
* Pregnant women are excluded from this study because gadolinium-based agents have not been proven to be safe to administer to a developing fetus. Similarly, breastfeeding women will be excluded from this study.
* Patients with a prior diagnosis of brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 214 (Estimated)
Dates: Start 2019-07-26 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Neurologic Quality of Life at 12 Months using the MD Anderson Symptom Inventory - Brain Tumor Module | 12 Months
  For patients with HR+/HER2- or HER2+ metastatic breast cancer
Incidence of Symptomatic Brain Metastases | Through study completion, an average of 1 year
  For patients with triple negative metastatic breast cancer
Incidence of Brain Metastases | Through study completion, an average of 1 year
  For patients with inflammatory breast cancer managed with curative intent

SECONDARY OUTCOMES:
Number of brain metastases | Through study completion, an average of 1 year
Size of brain metastases | Through study completion, an average of 1 year
Development of metastases in the brainstem as seen on magnetic resonance imaging of the brain | Through study completion, an average of 1 year
Development of leptomeningeal carcinomatosis as seen on magnetic resonance imaging of the brain | Through study completion, an average of 1 year
Radiographic appearance of brain metastases | Through study completion, an average of 1 year
Development of symptomatic brain metastases based on review of medical notes / history | Through study completion, an average of 1 year
Neurologic death | Through study completion, an average of 1 year
All-cause mortality | Through study completion, an average of 1 year
Development of seizures based on review of medical notes / history | Through study completion, an average of 1 year
Receipt of whole brain radiation due to brain metastases | Through study completion, an average of 1 year
Receipt of neurosurgical resection due to brain metastases | Through study completion, an average of 1 year
Quality of life assessment via EuroQol Group 5D Instrument | Through study completion, an average of 1 year
Neurocognitive function using the Hopkins Verbal Learning Test Instrument | Through study completion, an average of 1 year
Neurocognitive function using the Trail Making Test Instrument | Through study completion, an average of 1 year
Neurocognitive function using the Controlled Oral Word Association Test | Through study completion, an average of 1 year
Neurocognitive function using the Mini-Mental Status Exam Instrument | Through study completion, an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ayal Aizer, MD, MHS, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to: [contact information for Sponsor Investigator or designee]. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: BWH - Contact the Partners Innovations team at http://www.partners.org/innovation DFCI - Contact the Belfer Office for Dana-Farber Innovations (BODFI) at innovation@dfci.harvard.edu